CLINICAL TRIAL: NCT01810562
Title: Study on Effect of Tactile Stimulation on Reduced Sensibility of the Affected Extremities After Stroke.
Brief Title: SlagSens (Effect of Tactile Stimulation After Stroke)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not able to include enough participants.
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 4403 001
Record Dates: First submitted 2013-03-05; First posted 2013-03-13 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: Stroke; Tactile; Sensibility; Stimulation; Extremities; Arm; Leg
MeSH Terms: conditions — Stroke | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specific treatment + std stroke care (Experimental): Specific treatment in addition to standard stroke care
  Interventions: Other: Specific treatment in addition to standard stroke care
- Std stroke care (No Intervention): Patients receive only standard stroke treatment and no specific treatment.

INTERVENTIONS:
Other: Specific treatment in addition to standard stroke care — Stimulation of both the affected side and not affected side. Treatment twice per day for three months. Unperturbed side always stimulated first.
  Isstimulering achieved by an ice cube melted on each of the affected ektremitetene evenly distributed.
  Brushing on thin clothing or directly on the skin, 10 times rapidly for each location. On the back of m. deltoideus from right to left side of the body, laterally along the humerus, frontally, along the radius / ulna laterally, frontal and dorsal palm, along the femur first laterally and frontally, along the tibia / fibula laterally, frontally and the footplate dorsal side.
  Scrolling with spiked ball over the same area as brushing for two minutes evenly.
  Firm pressure for two minutes evenly in the same area.
  Other Names: Icestimulation; Firm pressure; Brushing with soft brush; Rolling with spiked ball
  Arms: Specific treatment + std stroke care

SUMMARY:
The purpose of this study is to determine whether tactile stimulation for reduced sensibility of the affected extremities after stroke has effect.

Hypothesis:

Stimulation of sensibility after stroke will have a significant contribution for improved sensibility. Without any stimulation, no signal is sent to the brain and there is no need for the healthy parts of the brain to adapt this function. Stimulation of the sensibility over a period of time on both sides of the body, gives the brain signals and the opportunity to compare how the signals should be recognized. New connection will be able to interpret signals correctly.

DETAILED DESCRIPTION:
Through stroke rehabilitation, function from damaged areas can be replaced by healthy parts of the brain. It is important for rehabilitation to take advantage of this compensatory qualities whit early intervention and mobilization. Only small gains can lead to big improvements.

About half of stroke survivors gets reduced sensibility caused bye the stroke, and sensibility is considered to be an important part of rehabilitation of function and activities.

A Norwegian guideline concludes that the scientific knowledge is to week to recommend this kind of treatment. There is some evidence for improvement of sensibility when specific training and stimulation is given. Achievements in sensibility can lead to some improvement in function.

The project will be carried out as a randomized controlled trial. In this project, the intervention group receive tactile senses stimulated twice daily over a period of 3 months, while the control group receives standard treatment. The results from both groups are measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with impaired tactile sensitivity after stroke Kongsberg hospital to undergo rehabilitation course.

Exclusion Criteria:

* Patients with a history of stroke.
* Patients with significant symptomatic additional diseases, such as neuropathy.
* Patients who cannot provide adequate response if they can feel the touch.
* Terminal and palliative care patients.
* Patients with cancer.
* Patients with hypertonic muscles in the current body area.
* Patients below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Weinstein Enhanced sensory test (WEST) | Change within 3 days after the patient has been hospitalized to 3 months
  Measurement of defined points on the arms and legs.

SECONDARY OUTCOMES:
Disk-Criminator | Change from 3 days after the patient has been hospitalized to 3 months
  Measurement of defined points on the arms and legs.
NIH Stroke Scale (NIHSS) | Change from Baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn A Graff, PhD, Study Director — Vestre Viken Hospital Trust; Bente Kristensen, BSc, Principal Investigator — Vestre Viken Hospital Trust
Locations (1):
- Vestre Viken Health, clinic Kongsberg Hostpital, Kongsberg, Buskerud, Norway